CLINICAL TRIAL: NCT06863493
Title: Study of the Safety and Effectiveness of Oral SFA-002 Compared to Oral Apremilast (Otezla) Tablets and Placebo in Mild to Severe Plaque Psoriasis
Brief Title: Comparison of Otezla to SFA-002 to Placebo in Plaque Psoriasis Patients
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SFA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFA-002-04
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis (PsO)
Keywords: Otezla; apremilast; Mild psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SFA002 (Experimental): SFA002 750mg 2 times daily
  Interventions: Drug: SFA002; Drug: Placebo
- Otezla (apremilast) (Experimental): 30mg 2 times daily
- Matched Placebo (Placebo Comparator)
  Interventions: Drug: SFA002; Drug: Placebo

INTERVENTIONS:
Drug: SFA002 — SFA002 760mg
  Arms: Matched Placebo; SFA002
Drug: Otezla — Oral Otezla 30mg
Drug: Placebo — Placebo will be matched to whichever drug is assigned when randomized
  Arms: Matched Placebo; SFA002

SUMMARY:
The goal of this clinical trial] is to learn if SFA002 can treat mild, moderate and severe plaque psoriasis as good or better than Otezla, compared to placebo in adult and pediatric patients.

The main questions it aims to answer are:

How much does oral SFA002 treatment improve plaque psoriasis measured at different timepoints, 12 weeks, 24 weeks and 52 weeks of treatment.

How much does Oral Otezla (Apremilast) improve plaque psoriasis measured at different timepoints, 12 weeks, 24 weeks and 52 weeks of treatment.

These treatments will be compared to placebo, a look-alike substance that contains no drug.

Participants will be randomly placed into 3 groups to receive either SFA002, or oral apremilast or placebo for the duration of the trial. Patients that do not respond to apremilast or placebo treatment in 12 weeks will be offered the opportunity to take SFA002 for the remainder of the study.

There may be a higher burden for participants in this study compared to usual standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:-

1. Candidates for systemic therapy with mild to moderate chronic plaque psoriasis (PsO) (with or without psoriatic arthritis) at Screening and Baseline for at least 6 months prior to Baseline defined as:
2. Body Surface Area (BSA) >= 10% and <= 15%; and Psoriasis Area and Severity Index (PASI) >= 12; and Static Physician Global Assessment (sPGA) = 3 (moderate) based on a 5-point scale (0 to 4) -

Exclusion Criteria:

1. Participant has any form of PsO other than chronic plaque PsO (e.g., pustular PsO, palmoplantar pustulosis, acrodermatitis of Hallopeau, erythrodermic, or guttate PsO).
2. History of current drug-induced PsO or a drug-induced exacerbation of pre-existing psoriasis.
3. History of active ongoing inflammatory skin diseases other than PsO and psoriatic arthritis that could interfere with the assessment of PsO (e.g., hyperkeratotic eczema).
4. Prior exposure to SFA002 or apremilast. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Psoriasis Area Severity Index (PASI) 90 (Defined as at Least 90% Improvement in PASI From Baseline) in Intent to Treat Population at Week 12 (ITT_A) | Week 12
  The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with higher scores indicating more severe disease.
Percentage of Participants Achieving Static Physician Global Assessment (sPGA) 0 or 1 With at Least 2-grade Improvement From Baseline in Intent to Treat Population at Week 12 (ITT_A) | 12 weeks
  The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions. Scores range from 0 (clear) to 4 (severe).
Percentage of Participants Achieving PASI 90 in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR) | week 52
  The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving PASI 75 (Defined as at Least 75% Improvement in PASI From Baseline) in Intent to Treat Population at Week 12 (ITT_A) | Week 12
  The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with higher scores indicating more severe disease.
Percentage of Participants Achieving PASI 75 in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR) | week 52
  The PASI is used to evaluate a participant's overall psoriasis disease state that includes the percent of surface area of skin that is affected and the severity of erythema, induration, and desquamation over four body regions (head, upper extremities, trunk, and lower extremities). Scores range from 0 to 72, with higher scores indicating more severe disease.
Percentage of Participants Achieving Static Physician Global Assessment (sPGA) 0 or 1 With at Least 2-grade Improvement From Baseline in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR) | Week 52
  Percentage of Participants Achieving Static Physician Global Assessment (sPGA) 0 or 1 With at Least 2-grade Improvement From Baseline in Intent to Treat Population for Apremilast Non-Responders at Week 52 (ITT_B_NR)

IPD SHARING:
Plan to Share IPD: Undecided